CLINICAL TRIAL: NCT03850275
Title: The Effects of E+Shots Energy Beverage on Mood, Cognitive Function, Heart Rate, Blood Pressure, and Fine Motor Task Performance
Brief Title: The Effects of e+Shots Energy Beverage on Mental Energy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clarkson University (Other)
Collaborators: Isagenix International LLC (Industry)
Responsible Party: Principal Investigator, Ali Boolani, Assistant Professor, Clarkson University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-05
Record Dates: First submitted 2018-07-18; First posted 2019-02-21 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Caffeine
MeSH Terms: interventions — Methods; Therapeutics

STUDY DESIGN:
Intervention Model Description: Crosover Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental: Placebo, then caffeinated placebo, then e+shots (Experimental): Participants received placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the caffeinated placebo and tested for 108 minutes. After another 48 hour washout period they received the e+shot and were tested for 108 minutes
  Interventions: Dietary Supplement: Intervention/treatment
- Experimental: Caffeinated placebo, then placebo, then e+shots (Experimental): Participants received caffeinated placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the placebo and tested for 108 minutes. After another 48 hour washout period they received the e+shot and were tested for 108 minutes
  Interventions: Dietary Supplement: Intervention/treatment
- Experimental: placebo, then e+shots, then caffeinated placebo (Experimental): Participants received placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received e+shots and tested for 108 minutes. After another 48 hour washout period they received the caffeinated placebo and were tested for 108 minutes.
  Interventions: Dietary Supplement: Intervention/treatment
- Experimental: caffeinated placebo, then e+shots, then placebo (Experimental): Participants received caffeinated placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the e+shots and tested for 108 minutes. After another 48 hour washout period they received the placebo and were tested for 108 minutes.
  Interventions: Dietary Supplement: Intervention/treatment
- Experimental: e+shots, then caffeinated placebo, then placebo (Experimental): Participants received e+shots and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the caffeinated placebo and tested for 108 minutes. After another 48 hour washout period they received the placebo and were tested for 108 minutes.
  Interventions: Dietary Supplement: Intervention/treatment
- Experimental: e+shots, then placebo, then caffeinated placebo (Experimental): Participants received e+shots and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the placebo and tested for 108 minutes. After another 48 hour washout period they received the caffeinated placebo and were tested for 108 minutes.
  Interventions: Dietary Supplement: Intervention/treatment

INTERVENTIONS:
Dietary Supplement: Intervention/treatment — Subjects received all 3 interventions Placebo ~3mg caffeine Caffeinated placebo ~100mg caffeine E+shots- The 4oz adaptogen-rich (E+shots) was E+ Shots (Isagenix International, LLC) containing approximately 90mg caffeine from green tea Camellia sinesis leaf extract (50%) and yerba maté extract (25%) along with a proprietary blend of adaptogenic herbs, including: eleutherococcus senticosus, crateagus oxycantha, rhodiola rosea and Schisandra chinensis.

SUMMARY:
The aim of the research project is to determine the changes in motivation to perform mental and physical tasks, feelings of vigor and fatigue, mental task vigilance and fine motor function after consumption of a commercially available energy product. The purpose of this study is determine whether e+shot, a product containing natural caffeine, will impact mood and performance up to 108 minutes post consumption compared to a sweetened solution containing synthetic caffeine.

DETAILED DESCRIPTION:
Enrolled participants who are low consumers of caffeine will be administered either a placebo (3mg caffeine), caffeinated placebo (~100mg of caffeine) or e+shot first and then will be crossed over to receive the other two interventions. The study consists of 3 treatment periods of 108 minutes each with a washout period of 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45
* Body Mass Index (BMI) < 30
* Profile of Mood Status Short Scale (POMS) score <13 on the energy scale
* Energy and Fatigue trait scale score <=10
* Consumption of <200mg of caffeine/day
* Consumption of <150 servings of polyphenols/month

Exclusion Criteria:

* Subjects taking prescription or over the counter medications (except for oral contraceptives) for a chronic medical condition or recreational drugs will be excluded Chronic medical conditions are any health condition that is expected to last more than 3 months and requires on going medical care such as coronary artery disease, multiple sclerosis, etc..
* Women who are pregnant or may be trying to become pregnant
* Women who are breastfeeding
* People who have been diagnosed with heart conditions and/or hypertension
* People who have liver disorders
* People who have sensitivity or allergy to caffeine
* People who have bipolar disorder
* People who have iron deficiency
* People who are allergic to plants of the Asteraceae/Compositae/Daisy family
* Day of testing

  * Subjects who have had a change of ±2 hours of sleep from their regular sleep time will be re-scheduled.
  * If subjects begin taking a prescription or over the counter medication for an acute condition (i.e. required to take the prescription or over the counter medication for < 3 months) during the study they will be given the option of continuing the study after they are no longer taking the prescription or over the counter medication or dropping out of the study.
  * If subjects are diagnosed with a chronic condition that requires the use of prescription medications for > 3 months after they have started the study they will be eliminated from the study.
  * Resting systolic BP > 180mmHg and diastolic BP > 90mmHg after consuming the caffeine beverage.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-26 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

IPD SHARING:
Plan to Share IPD: No
No plans to share individual participant data with other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After screening 1035 surveys, 30 participants completed the study (see Figure 1). Recruitment and data collection lasted from September 25th 2015 to December 10th, 2016 until 30 participants had completed all 3 days of treatment. There were no harms or unintended consequences for any of the interventions.
Pre-assignment Details: 43 participants were randomized. Of the 43 participants who were randomized, 13 did not start the study due to scheduling conflicts and were un-enrolled from the study.
Groups:
- Placebo, Then Caffeinated Placebo, Then e+Shots: Participants received the placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the caffeinated placebo and tested for 108 minutes. After another 48 hour washout period they received the e+shot and were tested for 108 minutes
- Placebo, Then e+Shots, Then Caffeine: Participants received the placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received e+shots and tested for 108 minutes. After another 48 hour washout period they received the caffeinated placebo and were tested for 108 minutes
- Caffeinated Placebo, Then Placebo, Then e+Shots: Participants received the caffeinated placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the placebo and tested for 108 minutes. After another 48 hour washout period they received the e+shot and were tested for 108 minutes
- Caffeinated Placebo, Then e+Shots, Then Placebo: Participants received the caffeinated placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the e+shots and tested for 108 minutes. After another 48 hour washout period they received the placebo and were tested for 108 minutes
- e+Shots, Then Placebo, Then Caffeinated Placebo: Participants received the e+shots and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the placebo and tested for 108 minutes. After another 48 hour washout period they received the placebo and were tested for 108 minutes
- e+Shots, Then Caffeinated Placebo, Then Placebo: Participants received the e+shots and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the caffeinated placebo and tested for 108 minutes. After another 48 hour washout period they received the placebo and were tested for 108 minutes
Period: Overall Study
Arm/Group | Placebo, Then Caffeinated Placebo, Then e+Shots | Placebo, Then e+Shots, Then Caffeine | Caffeinated Placebo, Then Placebo, Then e+Shots | Caffeinated Placebo, Then e+Shots, Then Placebo | e+Shots, Then Placebo, Then Caffeinated Placebo | e+Shots, Then Caffeinated Placebo, Then Placebo
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 30 participants received all 3 interventions.
Groups:
- Placebo, Then e+Shots, the Caffeinated Placebo: Participants received the placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the e+shots and tested for 108 minutes. After another 48 hour washout period they received the caffeinated placebo and were tested for 108 minutes
- Caffeinated Placebo, Then e+Shots, Then Placebo: Participants received the caffeinated placebo and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the e+shot and tested for 108 minutes. After another 48 hour washout period they received the placebo and were tested for 108 minutes
- E+Shots, Then Placebo, Then Caffeinated Placebo: Participants received the e+shot and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the placebo and tested for 108 minutes. After another 48 hour washout period they received the caffeinated placebo and were tested for 108 minutes
- E+Shot, Then Caffeinated Placebo, Then Placebo: Participants received the e+shot and were tested for 108 minutes after consumption. After a 48 hour washout period, they received the caffeinated placebo and tested for 108 minutes. After another 48 hour washout period they received the placebo and were tested for 108 minutes
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Caffeinated Placebo, Then e+Shots | Placebo, Then e+Shots, the Caffeinated Placebo | Caffeinated Placebo, Then Placebo, Then e+Shots | Caffeinated Placebo, Then e+Shots, Then Placebo | E+Shots, Then Placebo, Then Caffeinated Placebo | E+Shot, Then Caffeinated Placebo, Then Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (1.34) | 21.8 (5.85) | 22 (3.94) | 20 (1.87) | 20.4 (2.88) | 26 (6.89) | 21.8 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 3 | 2 | 3 | 17
  Male | 3 | 2 | 1 | 2 | 3 | 2 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 0 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 2 | 4
  White | 2 | 2 | 5 | 5 | 5 | 2 | 21
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 165.61 (15.28) | 164.59 (10.38) | 163.58 (8.91) | 164.59 (16.40) | 179.32 (6.86) | 174.75 (17.08) | 169.6 (12.4)
Weight [Mean (Standard Deviation); unit: kg] | 67.68 (9.47) | 67.27 (25.62) | 66.73 (12.48) | 67.18 (17.64) | 71.18 (7.58) | 74.91 (16.30) | 67.6 (11.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in POMS Vigor
Description: POMS Vigor, Scores range from 0-20 with higher scores indicating improved outcome
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: <3mg of caffeine
  Placebo: ~3mg caffeine
- Caffeinated Placebo: ~100mg caffeine
  Caffeinated placebo: ~100mg of synthetic caffeine
- E+Shots: ~100mg caffeine + adaptogens
  E+shots: The 4oz adaptogen-rich (E+shots) was E+ Shots (Isagenix International, LLC) containing approximately 90mg caffeine from green tea Camellia sinesis leaf extract (50%) and yerba maté extract (25%) along with a proprietary blend of adaptogenic herbs, including: eleutherococcus senticosus, crateagus oxycantha, rhodiola rosea and Schisandra chinensis.
Arm/Group | Placebo | Caffeinated Placebo | E+Shots
Number analyzed (Participants) | 30 | 30 | 30
score on a scale
  Pre-beverage-0 minutes | 9.03 (4.63) | 8.93 (4.60) | 8.80 (4.60)
  Post-beverage 1- 30 minutes | 9.03 (4.17) | 10.13 (3.91) | 9.67 (4.03)
  Post-beverage 2-68 minutes | 9.33 (4.33) | 9.87 (4.38) | 9.76 (4.27)
  Post-beverage 3-108 minutes | 9.38 (4.59) | 9.89 (5.22) | 10.15 (4.54)

2. Primary Outcome: Change in POMS Fatigue
Description: POMS Fatigue Scores range from 0-20with higher scores indicating worse outcome
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- E+Shot: ~100mg caffeine + adaptogens E+shots: The 4oz adaptogen-rich (E+shots) was E+ Shots (Isagenix International, LLC) containing approximately 90mg caffeine from green tea Camellia sinesis leaf extract (50%) and yerba maté extract (25%) along with a proprietary blend of adaptogenic herbs, including: eleutherococcus senticosus, crateagus oxycantha, rhodiola rosea and Schisandra chinensis.
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre-beverage- 0 minutes | 8.03 (2.94) | 8.00 (2.89) | 8.17 (2.81)
  Post -beverage 1-30 minutes | 8.13 (2.98) | 7.07 (2.48) | 7.67 (2.94)
  Post -beverage 2-68 minutes | 8.23 (2.62) | 7.66 (3.27) | 7.57 (2.81)
  Post-beverage 3-108 minutes | 7.72 (2.55) | 7.77 (3.15) | 8.07 (3.22)

3. Primary Outcome: Change in POMS Depression
Description: POMS Depression Scores range from 0-20 with higher scores indicating worse outcome
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre-beverage- 0 minutes | 5.37 (1.07) | 5.50 (1.41) | 5.30 (0.65)
  Post-beverage 1- 30 minutes | 5.43 (1.04) | 5.50 (1.20) | 5.23 (0.63)
  Post-beverage 2-68 minutes | 5.30 (0.84) | 5.45 (1.27) | 5.20 (0.61)
  Post-beverage 3-108 minutes | 5.28 (0.65) | 5.31 (1.01) | 5.25 (0.59)

4. Primary Outcome: Change in POMS Anxiety
Description: POMS Anxiety Scores range from 0-20 with higher scores indicating worse outcome
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre-beverage-0 minutes | 5.43 (0.73) | 5.63 (1.16) | 5.60 (1.30)
  Post-beverage 1- 30 minutes | 5.40 (0.77) | 5.73 (1.34) | 5.77 (1.28)
  Post-beverage 2-68 minutes | 5.40 (0.72) | 5.66 (1.52) | 5.87 (1.25)
  Post-beverage 3-108 minutes | 5.52 (0.91) | 5.62 (1.10) | 5.64 (1.03)

5. Primary Outcome: Change in POMS Anger
Description: POMS Anger Scores range from 0-20 with higher scores indicating worse outcome
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre-beverage-0 minutes | 5.27 (0.79) | 5.47 (0.71) | 5.90 (1.27)
  Post-beverage 1- 30 minutes | 5.30 (0.65) | 5.33 (0.71) | 5.53 (1.31)
  Post-beverage 2-68 minutes | 5.60 (1.04) | 5.41 (1.35) | 5.47 (0.94)
  Post-beverage 3-108 minutes | 5.31 (0.85) | 5.27 (0.53) | 5.57 (1.20)

6. Primary Outcome: Change in POMS Confusion
Description: POMS Anger Scores range from -4 to 16 with higher scores indicating worse outcome
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minute
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre-beverage-0 minutes | 2.50 (1.25) | 2.73 (1.57) | 2.70 (1.54)
  Post-beverage 1- 30 minutes | 2.57 (1.17) | 2.33 (1.45) | 2.17 (1.21)
  Post-beverage 2-68 minutes | 2.50 (1.04) | 2.59 (1.57) | 2.43 (1.43)
  Post-beverage 3-108 minutes | 2.34 (1.05) | 2.58 (1.60) | 2.29 (1.56)

7. Primary Outcome: Change in Serial Subtraction 3 Task Performance
Description: Serial subtraction 3- Number of attempts
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: attempts
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
attempts
  Pre-beverage-0 minutes | 46.23 (16.18) | 48.20 (14.59) | 46.27 (16.45)
  Post-beverage 1- 30 minutes | 52.77 (15.84) | 50.63 (15.90) | 54.86 (15.92)
  Post-beverage 2-68 minutes | 54.47 (16.11) | 53.50 (15.36) | 54.34 (16.32)
  Post-beverage 3-108 minutes | 56.10 (16.01) | 57.21 (15.98) | 55.33 (16.60)

8. Primary Outcome: Change in Serial Subtraction 3 Task Performance
Description: Serial subtraction 3- Number correct
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: correct attempts
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
correct attempts
  Pre-beverage-0 minutes | 44.80 (16.24) | 46.27 (14.70) | 44.23 (17.08)
  Post-beverage 1- 30 minutes | 51.17 (15.57) | 48.70 (16.08) | 52.97 (16.16)
  Post-beverage 2-68 minutes | 52.63 (16.26) | 51.37 (15.54) | 51.82 (16.91)
  Post-beverage 3-108 minutes | 53.38 (16.15) | 54.59 (16.90) | 52.17 (17.85)

9. Primary Outcome: Change in Serial Subtraction 3 Task Performance
Description: Serial subtraction 3- Percentage correct
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre-beverage-0 minutes | 96.35 (3.98) | 95.69 (4.23) | 94.43 (6.85)
  Post-beverage 1- 30 minutes | 96.98 (3.07) | 95.76 (3.69) | 96.22 (3.88)
  Post-beverage 2-68 minutes | 96.21 (3.18) | 95.57 (3.38) | 92.78 (7.83)
  Post-beverage 3-108 minutes | 95.09 (4.48) | 93.96 (8.89) | 93.79 (6.63)

10. Primary Outcome: Change in Serial Subtraction 7 Task Performance
Description: Serial subtraction 7- Number of attempts
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: attempts
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
attempts
  Pre-beverage-0 minutes | 26.53 (10.19) | 27.90 (10.13) | 28.77 (11.04)
  Post-beverage 1- 30 minutes | 29.38 (10.71) | 30.80 (11.25) | 32.60 (10.99)
  Post-beverage 2-68 minutes | 31.57 (12.09) | 33.07 (11.38) | 33.47 (11.60)
  Post-beverage 3-108 minutes | 33.90 (12.11) | 35.69 (12.02) | 34.27 (13.02)

11. Primary Outcome: Change in Serial Subtraction 7 Task Performance
Description: Serial subtraction 7- Number correct
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: correct attempts
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
correct attempts
  Pre-beverage-0 minutes | 24.73 (10.70) | 26.17 (10.30) | 27.00 (11.23)
  Post -beverage 1-30 minutes | 27.83 (10.70) | 29.03 (10.81) | 30.20 (10.95)
  Post-beverage 2-68 minutes | 28.83 (11.81) | 31.27 (11.59) | 30.41 (11.84)
  Post-beverage 3-108 minutes | 30.43 (11.43) | 33.48 (11.96) | 31.60 (13.15)

12. Primary Outcome: Change in Serial Subtraction 7 Task Performance
Description: Serial subtraction 7- Percentage correct
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre-beverage-0 minutes | 92.53 (8.80) | 92.78 (7.99) | 92.72 (11.29)
  Post-beverage 1- 30 minutes | 94.36 (4.98) | 93.59 (8.08) | 91.65 (8.13)
  Post-beverage 2-68 minutes | 92.92 (8.42) | 93.80 (6.60) | 91.44 (7.21)
  Post-beverage 3-108 minutes | 91.21 (8.74) | 93.17 (6.07) | 90.60 (9.18)

13. Primary Outcome: Change in Blood Pressure
Description: Blood pressure- systolic and diastolic measured in mmHg
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo Systolic; Placebo Diastolic: <3mg of caffeine Placebo: ~3mg caffeine
- E+Shot Systolic; E+Shot Diastolic: ~100mg caffeine + adaptogens E+shots: The 4oz adaptogen-rich (E+shots) was E+ Shots (Isagenix International, LLC) containing approximately 90mg caffeine from green tea Camellia sinesis leaf extract (50%) and yerba maté extract (25%) along with a proprietary blend of adaptogenic herbs, including: eleutherococcus senticosus, crateagus oxycantha, rhodiola rosea and Schisandra chinensis.
- Caffeinated Placebo Systolic; Caffeinated Placebo Diastolic: ~100mg caffeine Caffeinated placebo: ~100mg of synthetic caffeine
Arm/Group | Placebo Systolic | Placebo Diastolic | E+Shot Systolic | E+Shot Diastolic | Caffeinated Placebo Systolic | Caffeinated Placebo Diastolic
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30
mmHg
  Pre-beverage-0 minutes | 111.80 (12.22) | 71.00 (8.51) | 111.00 (16.18) | 71.50 (9.44) | 109.63 (12.99) | 68.97 (9.04)
  Post-beverage 1- 30 minutes | 109.53 (12.62) | 71.30 (8.12) | 113.60 (13.74) | 72.30 (7.91) | 114.93 (16.41) | 74.07 (7.70)
  Post-beverage 2-68 minutes | 111.30 (15.50) | 73.60 (12.14) | 114.57 (16.45) | 74.80 (17.78) | 113.40 (15.07) | 74.37 (8.20)
  Post-beverage 3-108 minutes | 112.30 (13.37) | 72.57 (8.02) | 114.67 (14.21) | 72.03 (10.32) | 112.80 (15.04) | 73.17 (8.45)

14. Primary Outcome: Change in Heart Rate
Description: Heart rate- beats per minute
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
BPM
  Pre-beverage-0 minutes | 72.50 (13.86) | 70.13 (1.84) | 69.80 (13.99)
  Post-beverage 1- 30 minutes | 70.10 (13.98) | 65.23 (11.31) | 67.37 (12.35)
  Post-beverage 2-68 minutes | 68.00 (13.86) | 67.90 (14.51) | 67.10 (13.33)
  Post-beverage 3-108 minutes | 66.83 (14.18) | 64.47 (13.64) | 63.83 (12.36)

15. Primary Outcome: Change in Fine Motor Task Performance
Description: 9-hole peg test- measured in seconds- The validated nine-hole peg test of finger dexterity was used to measure fine motor control. The 12 cm × 12 cm wooden pegboard contained nine holes and was placed on the desktop in front of the seated participant. There were nine 0.64 cm wide cylindrical pegs, were placed on the desktop outside of the container on the right side of the board and on the left side of the board for when the participant's right hand and left hand were tested, respectively. Participants were instructed to place one peg at a time into the pegboard holes until they were filled, and then remove each peg one at a time onto the desktop as fast as they could, first with their dominant hand and next with their non-dominant hand. Each test was performed twice.
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Placebo Non-dominant Hand; Placebo Dominant Hand: <3mg of caffeine Placebo: ~3mg caffeine
- E+Shot Non-dominant Hand; E+Shot Dominant Hand: ~100mg caffeine + adaptogens E+shots: The 4oz adaptogen-rich (E+shots) was E+ Shots (Isagenix International, LLC) containing approximately 90mg caffeine from green tea Camellia sinesis leaf extract (50%) and yerba maté extract (25%) along with a proprietary blend of adaptogenic herbs, including: eleutherococcus senticosus, crateagus oxycantha, rhodiola rosea and Schisandra chinensis.
- Caffeinated Placebo Non-Dominant Hand; Caffeinated Placebo Dominant Hand: ~100mg caffeine Caffeinated placebo: ~100mg of synthetic caffeine
Arm/Group | Placebo Non-dominant Hand | Placebo Dominant Hand | E+Shot Non-dominant Hand | E+Shot Dominant Hand | Caffeinated Placebo Non-Dominant Hand | Caffeinated Placebo Dominant Hand
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30
Seconds
  Pre-beverage-0 minutes | 19.42 (2.94) | 18.87 (2.64) | 19.27 (2.65) | 18.60 (2.45) | 19.31 (3.40) | 18.65 (2.93)
  Post-beverage 1- 30 minutes | 18.80 (2.45) | 18.21 (2.50) | 18.88 (2.83) | 17.93 (2.09) | 18.73 (3.23) | 17.95 (2.79)
  Post-beverage 2-68 minutes | 18.70 (2.76) | 18.22 (2.86) | 18.58 (2.55) | 17.68 (12.07) | 18.78 (3.38) | 18.02 (2.95)
  Post-beverage 3-108 minutes | 18.54 (2.94) | 17.86 (2.75) | 18.17 (2.93) | 17.50 (2.20) | 18.44 (3.37) | 17.56 (2.84)

16. Primary Outcome: Change in State Mental Energy
Description: State Mental Energy- scores range from 0 to 300 with higher scores indicating better outcome
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre-beverage-0 minutes | 9.93 (6.01) | 10.27 (6.26) | 10.13 (7.39)
  Post-beverage 1- 30 minutes | 9.23 (6.30) | 8.70 (6.51) | 9.43 (7.23)
  Post-beverage 2-68 minutes | 9.90 (6.38) | 9.17 (6.66) | 9.52 (7.16)
  Post-beverage 3-108 minutes | 8.83 (5.42) | 9.73 (6.75) | 10.16 (7.71)

17. Primary Outcome: Change in State Physical Energy
Description: State Physical Energy- scores range from 0 to 300 with higher scores indicating better outcome
Time Frame: pre-beverage-0 minutes, Post beverage 1-30 minutes, Post beverage 2-68 minutes, Post beverage 3 -108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre beverage-0 minutes | 9.13 (5.87) | 9.50 (6.55) | 8.67 (6.14)
  Post 1 beverage-30 minutes | 8.43 (5.55) | 7.93 (6.11) | 8.67 (6.23)
  Post 2 beverage- 60 minutes | 8.63 (5.37) | 8.62 (6.38) | 8.83 (6.05)
  Post 3 beverage-108 minutes | 8.31 (5.55) | 8.37 (5.84) | 8.84 (6.58)

18. Primary Outcome: Change in State Mental Fatigue
Description: State mental fatigue- scores range from 0 to 300 with higher scores indicating worse outcome
Time Frame: pre beverage-0 minutes, post beverage 1- 30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre beverage- 0 minutes | 13.27 (6.59) | 13.40 (6.75) | 15.13 (6.58)
  Post 1 beverage-30 minutes | 13.30 (6.20) | 14.60 (7.12) | 15.60 (7.31)
  Post 2 beverage- 60 minutes | 13.67 (6.77) | 14.07 (7.10) | 15.34 (7.49)
  Post 3 beverage- 108 minutes | 13.90 (7.39) | 14.46 (7.12) | 16.44 (8.30)

19. Primary Outcome: Change in State Physical Fatigue
Description: State physical fatigue- scores range from 0 to 300 with higher scores indicating worse outcome
Time Frame: pre beverage-0, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Score on a scale
  Pre beverage-0 minutes | 13.87 (6.34) | 14.63 (15.97) | 16.40 (6.89)
  Post 1 beverage-30 minutes | 14.23 (6.35) | 15.37 (6.56) | 16.40 (7.38)
  Post 2 beverage- 60 minutes | 14.57 (6.36) | 15.31 (6.56) | 16.38 (7.27)
  Post 3 beverage- 108 minutes | 14.69 (6.89) | 15.31 (6.63) | 16.92 (7.24)

20. Primary Outcome: Change in Continuous Performance Task Performance Percent Correct
Description: Continuous Performance Task- Percentage of correct responses Participants monitored a continuous series of letters (A-Z; Tahoma Regular font, size 20 pt) presented on the screen for 1000 ms. Participants were told to respond to the detection of the letter "X" only when it was preceded by the letter "A" by striking the left key on the key pad. The task was scored for percentage of target strings correctly detected, errors of omission (missed targets), average reaction time for correct detections, and the number of false alarms. The task lasted for two minutes and 48 targets were randomly presented
Time Frame: pre beverage-0 minutes, post beverage 1- 30 minutes, post beverage 2- 68, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 83.92 (25.53) | 80.46 (29.50) | 84.93 (17.69)
  Post 1 beverage-30 minutes | 77.79 (25.49) | 78.18 (27.49) | 83.32 (21.01)
  Post 2 beverage- 60 minutes | 79.07 (23.83) | 82.95 (27.88) | 85.26 (22.34)
  Post 3 beverage- 108 minutes | 79.07 (23.83) | 86.40 (16.47) | 85.56 (14.23)

21. Primary Outcome: Change in Continuous Performance Task Performance Number Incorrect
Description: Continuous Performance Task- Number of incorrect responses
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage- 0 minutes | 0.44 (0.51) | 0.49 (0.79) | 0.44 (0.58)
  Post 1 beverage-30 minutes | 0.48 (0.48) | 0.59 (0.80) | 0.45 (0.71)
  Post 2 beverage- 60 minutes | 0.37 (0.82) | 0.51 (1.13) | 0.56 (0.78)
  Post 3 beverage- 108 minutes | 0.48 (0.74) | 0.41 (0.58) | 0.37 (0.63)

22. Primary Outcome: Change in Continuous Performance Task Performance Missed Responses
Description: Continuous Performance Task- Percentage of missed responses
Time Frame: pre beverage-0 minutes, post beverage 1- 30 minutes, post beverage 2- 68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 16.08 (25.53) | 19.54 (29.50) | 14.97 (17.36)
  Post 1 beverage-30 minutes | 22.21 (24.49) | 21.81 (27.49) | 16.68 (21.01)
  Post 2 beverage- 60 minutes | 20.21 (23.72) | 17.05 (27.88) | 14.73 (22.34)
  Post 3 beverage- 108 minutes | 20.91 (24.73) | 13.60 (16.47) | 14.44 (14.23)

23. Primary Outcome: Change in Continuous Performance Task Performance Reaction Time Correct Responses
Description: Continuous Performance Task- reaction time for correct responses
Time Frame: pre beverage-0 minutes, post beverage 1- 30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
ms
  Pre beverage-0 minutes | 1441.63 (304.19) | 1475.20 (76.56) | 1499.64 (102.77)
  Post 1 beverage-30 minutes | 1515.54 (95.82) | 157.81 (158.49) | 1495.55 (85.77)
  Post 2 beverage- 60 minutes | 1516.12 (111.05) | 1506.42 (91.91) | 1527.74 (122.18)
  Post 3 beverage- 108 minutes | 1498.28 (72.03) | 1525.09 (82.97) | 1474.22 (75.06)

24. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Primary Task Percentage Correct
Description: Rapid Visual Input Processing task- Primary task- percentage correct
Time Frame: pre beverage- 0 minutes, post beverage 1- 30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutese | 59.45 (24.98) | 60.78 (26.18) | 57.18 (27.66)
  Post 1 beverage-30 minutes | 61.79 (25.86) | 67.16 (23.99) | 64.70 (25.18)
  Post 2 beverage- 60 minutes | 65.18 (20.86) | 70.27 (24.57) | 67.13 (24.75)
  Post 3 beverage- 108 minutes | 62.52 (26.73) | 64.65 (20.36) | 71.38 (19.06)

25. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Primary Task Percent Missed
Description: Rapid Visual Input Processing task- Primary task- percentage missed
Time Frame: pre beverage-0 minutes, post beverage 1- 30 minutes, post beverage 2-68 minutes, post beverage 3- 108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 31.85 (22.01) | 29.82 (20.67) | 34.13 (24.30)
  Post 1 beverage-30 minutes | 28.65 (24.00) | 39.62 (25.39) | 28.85 (25.07)
  Post 2 beverage- 60 minutes | 27.43 (19.29) | 22.82 (20.58) | 20.51 (16.77)
  Post 3 beverage- 108 minutes | 30.73 (26.00) | 27.90 (19.70) | 20.69 (17.00)

26. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Primary Task Incorrect Responses
Description: Rapid Visual Input Processing task- Primary task- incorrect responses
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 8.70 (9.57) | 9.40 (9.64) | 8.65 (10.28)
  Post 1 beverage-30 minutes | 9.55 (8.72) | 6.58 (8.34) | 6.50 (7.30)
  Post 2 beverage- 60 minutes | 7.33 (8.27) | 6.47 (8.96) | 9.88 (10.50)
  Post 3 beverage- 108 minutes | 7.33 (8.27) | 7.27 (5.79) | 7.54 (7.88)

27. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Primary Task Reaction Time for Percent Correct
Description: Rapid Visual Input Processing task- Primary task- reaction time for percent correct
Time Frame: pre beverage- 0 minutes, post beverage 1-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
ms
  Pre beverage-0 minutes | 777.76 (93.09) | 782.84 (99.82) | 786.74 (121.13)
  Post 1 beverage-30 minutes | 761.51 (74.29) | 774.57 (71.21) | 773.95 (75.76)
  Post 2 beverage- 60 minutes | 791.83 (55.05) | 752.33 (85.85) | 73.10 (76.58)
  Post 3 beverage- 108 minutes | 770.84 (71.41) | 736.22 (49.30) | 727.96 (79.60)

28. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Secondary Task Percent Correct
Description: Rapid Visual Input Processing task- Secondary task- percentage correct
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 58.75 (21.45) | 55.24 (23.10) | 55.28 (58.93)
  Post 1 beverage-30 minutes | 54.75 (19.69) | 59.98 (25.75) | 58.93 (27.25)
  Post 2 beverage- 60 minutes | 54.32 (24.46) | 57.05 (30.08) | 58.56 (28.20)
  Post 3 beverage- 108 minutes | 61.11 (24.75) | 61.56 (23.46) | 63.98 (24.26)

29. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Secondary Task Percentage Missed Responses
Description: Rapid Visual Input Processing task- Secondary task- percentage missed responses
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 39.85 (20.24) | 42.08 (22.55) | 43.64 (24.28)
  Post 1 beverage-30 minutes | 44.42 (19.59) | 39.62 (25.39) | 41.07 (27.25)
  Post 2 beverage- 60 minutes | 45.17 (24.55) | 0.42 (29.88) | 41.07 (28.36)
  Post 3 beverage- 108 minutes | 38.28 (24.45) | 37.35 (22.83) | 35.63 (24.38)

30. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Secondary Task Incorrect Responses
Description: Rapid Visual Input Processing task- Secondary task- incorrect responses
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2- 68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 1.36 (3.19) | 2.64 (5.37) | 1.09 (3.81)
  Post 1 beverage-30 minutes | 0.42 (1.86) | 0.00 (0.00) | 0.00 (0.00)
  Post 2 beverage- 60 minutes | 0.46 (1.96) | 0.83 (2.56) | 0.36 (1.71)
  Post 3 beverage- 108 minutes | 0.52 (2.08) | 1.04 (2.85) | 0.38 (1.78)

31. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Secondary Task Reaction Time for Correct Responses
Description: Rapid Visual Input Processing task- Secondary task- reaction time for correct responses
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
ms
  Pre beverage-0 minutes | 610.31 (124.82) | 66.66 (98.86) | 612.76 (65.11)
  Post 1 beverage-30 minutes | 627.79 (59.08) | 601.89 (76.14) | 604.52 (87.25)
  Post 2 beverage- 60 minutes | 628.47 (108.98) | 634.83 (102.15) | 621.75 (129.66)
  Post 3 beverage- 108 minutes | 649.46 (90.90) | 633.80 (67.24) | 598.90 (92.00)

32. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Tertiary Task Percentage Correct Responses
Description: Rapid Visual Input Processing task- Tertiary task- percentage correct responses
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 83.76 (19.05) | 88.89 (12.38) | 86.45 (11.74)
  Post 1 beverage-30 minutes | 84.05 (15.79) | 88.21 (14.81) | 90.61 (8.10)
  Post 2 beverage- 60 minutes | 85.57 (13.61) | 87.77 (16.48) | 85.90 (16.46)
  Post 3 beverage- 108 minutes | 88.09 (12.85) | 88.73 (14.23) | 89.59 (10.67)

33. Primary Outcome: Change in Rapid Visual Input Processing Task Performance- Tertiary Task Percent Missed Responses
Description: Rapid Visual Input Processing task- Tertiary task- percentage missed responses
Time Frame: pre beverage-0 minute, post beverage-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 12.56 (16.49) | 9.55 (11.72) | 11.18 (10.17)
  Post 1 beverage-30 minutes | 15.32 (15.85) | 10.30 (14.14) | 9.20 (11.32)
  Post 2 beverage- 60 minutes | 11.47 (11.41) | 11.40 (16.71) | 12.43 (15.63)
  Post 3 beverage- 108 minutes | 10.16 (13.55) | 8.42 (13.00) | 9.41 (10.60)

34. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Tertiary Task Number of Incorrect Responses
Description: Rapid Visual Input Processing task- Tertiary task- number of incorrect responses
Time Frame: pre beverage-0 minutes, post beverage 1- 30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
Percentage
  Pre beverage-0 minutes | 4.68 (7.09) | 3.10 (5.36) | 2.40 (4.55)
  Post 1 beverage-30 minutes | 2.57 (3.97) | 1.81 (4.35) | 2.98 (8.17)
  Post 2 beverage- 60 minutes | 3.05 (7.95) | 1.62 (3.42) | 3.07 (4.89)
  Post 3 beverage- 108 minutes | 2.92 (5.03) | 1.94 (3.61) | 1.52 (4.18)

35. Primary Outcome: Change in Rapid Visual Input Processing Task Performance Tertiary Task Reaction Time for Correct Responses
Description: Rapid Visual Input Processing task- Tertiary task- reaction time for correct responses
Time Frame: pre beverage-0 minutes, post beverage 1-30 minutes, post beverage 2-68 minutes, post beverage 3-108 minutes
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | E+Shot | Caffeinated Placebo
Number analyzed (Participants) | 30 | 30 | 30
ms
  Pre beverage-0 minutes | 749.10 (56.08) | 761.78 (60.50) | 752.61 (61.42)
  Post 1 beverage-30 minutes | 745.10 (61.10) | 731.21 (44.10) | 746.90 (53.46)
  Post 2 beverage- 60 minutes | 738.66 (56.00) | 728.52 (46.69) | 751.04 (55.61)
  Post 3 beverage- 108 minutes | 717.86 (40.95) | 737.23 (49.38) | 739.53 (58.21)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 141 minutes after beverage consumption
Description: No adverse events were reported
Arm/Group | Placebo | Caffeinated Placebo | E+Shots
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
There were technical problems with the Continuous Performance Task and Rapid Visual Input Processing task and not all data were interpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03850275/Prot_SAP_ICF_001.pdf